CLINICAL TRIAL: NCT06742931
Title: Discontinuation of Antiplatelet Agent After Drug-Coated Balloon Angioplasty in Stabilized Patients With High Bleeding Risk and Coronary Artery Disease
Brief Title: Drug-Coated Balloon Versus Drug-Eluting Stent for Treatment of De-Novo Coronary Lesions in Patients With High Bleeding Risk-2
Acronym: DCB-HBR-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Joo Myung Lee, Associate Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCT314316452025
Record Dates: First submitted 2024-12-15; First posted 2024-12-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Chronic Coronary Syndrome
Keywords: Coronary artery stenosis; Antiplatelet agent; Drug-coated balloon; Chronic coronary syndrome; Prognosis
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Intervention Model Description: A prospective, multi-center, open-label, randomized controlled, and superiority trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Clinical outcome assessment will be performed under blinded assessment about the allocated treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discontinuation of antiplatelet agent group (Experimental): In this group, antiplatelet monotherapy will be discontinued at the time of randomization. Randomization will be performed at 1 year from the index procedure using DCB angioplasty, standard duration of DAPT (1-3 months), and maintenance of antiplatelet monotherapy at least 1 year from the index procedure in patients with HBR and chronic coronary syndrome. In patients who are still under DAPT at 1 year from index DCB angioplasty, all antiplatelet agents will be discontinued after randomization.
  Interventions: Other: Discontinuation of antiplatelet agent group
- Continuation of antiplatelet agent group (Active Comparator): In this group, lifelong antiplatelet monotherapy will be continued after the time of randomization. Randomization will be performed at 1 year from the index procedure using DCB angioplasty, standard duration of DAPT (1-3 months), and maintenance of antiplatelet monotherapy at least 1 year from the index procedure in patients with HBR and chronic coronary syndrome. In patients who are still under DAPT at 1 year from index DCB angioplasty, DAPT will be changed to single antiplatelet therapy (aspirin or clopidogrel). The choice between aspirin or clopidogrel will be determined by the physician's discretion.
  Interventions: Other: Continuation of antiplatelet agent group

INTERVENTIONS:
Other: Discontinuation of antiplatelet agent group — In this group, antiplatelet monotherapy will be discontinued at the time of randomization. Randomization will be performed at 1 year from the index procedure using DCB angioplasty, standard duration of DAPT (1-3 months), and maintenance of antiplatelet monotherapy at least 1 year from the index procedure in patients with HBR and chronic coronary syndrome. In patients who are still under DAPT at 1 year from index DCB angioplasty, all antiplatelet agents will be discontinued after randomization.
  Arms: Discontinuation of antiplatelet agent group
Other: Continuation of antiplatelet agent group — In this group, lifelong antiplatelet monotherapy will be continued after the time of randomization. Randomization will be performed at 1 year from the index procedure using DCB angioplasty, standard duration of DAPT (1-3 months), and maintenance of antiplatelet monotherapy at least 1 year from the index procedure in patients with HBR and chronic coronary syndrome. In patients who are still under DAPT at 1 year from index DCB angioplasty, DAPT will be changed to single antiplatelet therapy (aspirin or clopidogrel). The choice between aspirin or clopidogrel will be determined by the physician's discretion.
  Arms: Continuation of antiplatelet agent group

SUMMARY:
A prospective, multi-center, open-label, randomized controlled, and superiority trial. The trial will compare clinical outcomes between discontinuation of antiplatelet agent and continuation of antiplatelet agent in HBR patients with chronic coronary syndrome treated by DCB angioplasty and standard duration of DAPT, followed by maintenance of single antiplatelet agent without clinical event for at least 1 year from the index procedure.

DETAILED DESCRIPTION:
In patients with chronic coronary syndrome, the benefit of percutaneous coronary intervention (PCI) has been controversial for a survival benefit while reducing the risk of spontaneous myocardial infarction (MI) or anginal symptoms. Therefore, unlike patients with acute coronary syndrome, routine PCI with drug-eluting stents (DES) for patients with chronic coronary syndrome should be individualized, considering the risk of long term possibility of stent failure and the need for maintaining dual antiplatelet therapy (DAPT) for certain period due to permanent vascular implant and increased risk of bleeding, especially in patients with high bleeding risk (HBR). Drug-coated balloon (DCB), a novel treatment strategy, which has benefit of having shorter antiplatelet therapy duration due to the absence of metallic scaffolds and polymers, could be an alternative treatment for patients with chronic coronary syndrome, especially in patients with HBR. Given the expanding indications for DCB including de novo coronary artery lesions, shorter duration of DAPT, and potentially reduced risk of bleeding might be a reasonable treatment strategy in patients with HBR.

In current guidelines, standard duration of DAPT after PCI is recommended for 1 to 3 months in patients with HBR. Then, it is recommended as Class IA recommendation for maintaining single antiplatelet agent for lifelong as a secondary prevention, regardless of the devices used during PCI and the risk of patients' bleeding risk. However, it should be noted that the supporting evidence for lifelong maintenance of single antiplatelet agent were derived from previous randomized controlled trials conducted in patients with acute myocardial infarction or stroke. In addition, the supporting evidence for lifelong maintenance of single antiplatelet agent after PCI was derived from the recent randomized controlled trials using metallic stents including bare metal stent, 1st generation DES, or 2nd generation DES. The gap in the evidence is that no previous trial evaluated the need of lifelong maintenance of single antiplatelet agent in HBR patients with chronic coronary syndrome treated by DCB angioplasty after standard duration of DAPT. Furthermore, although recent trial have shown that long-term antiplatelet monotherapy with clopidogrel demonstrated better clinical outcomes than antiplatelet monotherapy with aspirin in patients with chronic coronary syndrome undergoing PCI with DES, there has been scarce data regarding long-term antiplatelet therapy for HBR patients with chronic coronary syndrome treated by DCB angioplasty after standard duration of DAPT.

On this background, the current trial aims to compare clinical outcomes between discontinuation of antiplatelet agent and continuation of antiplatelet agent in HBR patients with chronic coronary syndrome treated by DCB angioplasty and standard duration of DAPT, followed by maintenance of single antiplatelet agent without clinical event for at least 1 year from the index procedure. Having this evidence will be able to more establish the evidence for the post-adjunctive medical treatment in patients with HBR after DCB angioplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 19 years of age
2. Subject who is able to understand risks, benefits and treatment alternatives and sign informed consent voluntarily.
3. Patients with chronic coronary syndrome and at least one de novo lesion of reference vessel size ≥2.25 mm, treated with DCB angioplasty
4. Patients with high bleeding risk: one or more of the criteria listed A. Age ≥ 75 years old B. Baseline Hemoglobin <11 g/dl (or anemia requiring transfusion during the 4 weeks prior to randomization) C. Any prior intra-cerebral bleed D. Hospital admission for bleeding during the prior 12 months E. Non skin cancer diagnosed or treated < 3 years F. Planned daily NSAID (other than aspirin) or steroids for >30 days after PCI G. Planned surgery that would require interruption of DAPT (within next 12 months) H. Renal failure defined as calculated creatinine clearance <40 ml/min or on dialysis I. Hematological disorders (platelet count <100,000/mm3 or any coagulation disorder) J. Severe chronic liver disease defined as patients who have developed any of the following: variceal hemorrhage, ascites, hepatic encephalopathy or jaundice K. Expected non-compliance to secondary prevention medications after PCI for other medical reasons
5. Patients who completed standard duration of DAPT (1-3months) and followed by maintenance of single antiplatelet agent (aspirin or P2Y12 inhibitor) for at least 1 year from index procedure.
6. No bleeding (BARC 2, 3, or 5 bleeding) or ischemic events (cardiovascular death, non-fatal MI, or clinically-indicated repeat revascularization) for at least 1 year from index procedure.

Exclusion Criteria:

1. Patients unable to provide consent
2. Patients with acute myocardial infarction or unstable angina
3. Patients with known intolerance to aspirin, P2Y12 inhibitors, or components of DCB
4. Patients with indication of oral anticoagulant
5. Patients with concomitant drug-eluting stent implantation during index PCI
6. Patients with history of ischemic stroke or previous myocardial infarction
7. Patients with peripheral arterial occlusive disease
8. Patients with angiographic findings of A. Left main coronary artery disease B. In-stent restenosis is the cause of target lesion C. Target lesion in bypass graft D. True bifurcation lesion that requires upfront 2-stenting E. Patients with residual stenosis on non-target vessels after PCI (>70% diameter stenosis or FFR≤0.80)
9. Patients who have non-cardiac co-morbid conditions with life expectancy <1 year
10. Patients who may result in protocol non-compliance (site investigator's medical judgment)
11. Patients with cardiogenic shock or cardiac arrest
12. Patients with severe left ventricular systolic dysfunction (ejection fraction <30%)
13. Patients with severe valvular heart disease requiring open heart surgery
14. Pregnant or lactating women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Major bleeding (BARC 2, 3, or 5 bleeding) | 1 year after last patient enrollment
  BARC 2, 3, or 5 bleeding

SECONDARY OUTCOMES:
Patient-oriented composite outcome | 1 year after last patient enrollment
  a composite of all-cause death, non-fatal myocardial infarction, and any revascularization
Cardiovascular death | 1 year after last patient enrollment
  Cardiovascular death
All-cause death | 1 year after last patient enrollment
  All-cause death
Target-vessel myocardial infarction | 1 year after last patient enrollment
  Target-vessel myocardial infarction
Non-fatal MI | 1 year after last patient enrollment
  Non-fatal MI
Clinically indicated target-lesion revascularization (TLR) | 1 year after last patient enrollment
  Clinically indicated target-lesion revascularization (TLR)
Clinically indicated target-vessel revascularization (TVR) | 1 year after last patient enrollment
  Clinically indicated target-vessel revascularization (TVR)
Any revascularization | 1 year after last patient enrollment
  Any revascularization
Cardiovascular death or target-vessel MI | 1 year after last patient enrollment
  Cardiovascular death or target-vessel MI
All-cause death or non-fatal MI | 1 year after last patient enrollment
  All-cause death or non-fatal MI
Target vessel failure | 1 year after last patient enrollment
  a composite of cardiovascular death, target-vessel MI, and clinically indicated target-vessel revascularization
Severe major bleeding (BARC 3 or 5 bleeding) | 1 year after last patient enrollment
  BARC 3 or 5 bleeding
Major bleeding (TIMI major bleeding) | 1 year after last patient enrollment
  TIMI major bleeding
Cerebrovascular accident (CVA) | 1 year after last patient enrollment
  Cerebrovascular accident (CVA) including Ischemic stroke, Hemorrhagic stroke, or Transient ischemic attack (TIA)

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Yong Hahn, MD, PhD, Study Chair — Samsung Medical Center; Young Bin Song, MD, PhD, Study Chair — Samsung Medical Center; Joo Myung Lee, MD, MPH, PhD, Principal Investigator — Samsung Medical Center
Locations (18):
- South Korea (18):
  - Korea University Ansan Hospital, Ansan
  - Keimyung University Dongsan Medical Center, Daegu
  - Gangneung Asan Hospital, University of Ulsan College of Medicine, Gangneung
  - Ilsan Paik hospital, Goyang
  - Chonnam National University Hospital, Chonnam National University Medical School, Gwangju
  - Chung-Ang University Gwangmyeong Hospital, Gwangmyeong
  - Catholic Kwandong University International St. Mary's Hospital, Incheon
  - Gachon Cardiovascular Research Institute, Gachon University, Incheon
  - Inha University Hospital, Incheon
  - Chonbuk National University Hospital and Chonbuk National University Medical School, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Chung-Ang University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Ajou University School of Medicine, Suwon
  - Uijeongbu St. Mary Hospital, Uijeongbu-si

IPD SHARING:
Plan to Share IPD: Yes
After completion of primary trial report, executive committee members will have discussion about sharing the individual participant data (IPD) upon reasonable requests,
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After completion of primary trial report
Access Criteria: Upon reasonable requests, executive committee members will have discussion about sharing the individual participant data (IPD).